CLINICAL TRIAL: NCT02868723
Title: PROspective Study to OPTimize thE HEALTH of Patients With TIAS (Transient Ischemic Attack) and Stroke Admitted to the Hamad General Hospital
Brief Title: PROspective Study to OPTimize thE HEALTH of Patients With TIAs (Transient Ischemic Attacks) and Stroke Admitted to the Hamad General Hospital
Acronym: PROMOTE-HEALTH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MRC-IRGC-02-NI-059
Record Dates: First submitted 2016-06-30; First posted 2016-08-16 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-08

CONDITIONS: Stroke; Transient Ischemic Attack (TIA)
Keywords: cerebrovascular disease; patient management; stroke management; prognosis; 3D Carotid Doppler Imaging; Randomization
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient; Cerebrovascular Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control; standard of care (No Intervention): All the subjects enrolled in this arm will receive counseling as the usual standard of care by the stroke neurologists. These will include procedures and guidelines as approved by American Heart Association (AHA), follow up and guidance as offered by Hamad General Hospital's policies.
- Intervention; Lifestyle counselling: Behavioural (Active Comparator): Subjects in this group will receive a more detailed guidance on rigorous management of stroke and will be provided assistance from a stroke trained nurse and pharmacist additional to the counseling offered by the Stroke Neurologist.
  Interventions: Other: Aggressive Management

INTERVENTIONS:
Other: Aggressive Management — With the aid of the nurse and pharmacist, the individuals in the interventional group will receive additional management of stroke by change is diet plan, increased exercise
  Arms: Intervention; Lifestyle counselling: Behavioural

SUMMARY:
This will be a prospective randomized 2 year study of patients admitted to the Hamad General Hospital (HGH) and the Stroke Prevention Clinic with a diagnosis of ischemic stroke (IS) and Transit ischemic attacks (TIAs). After signing of the informed consent forms and initial evaluation and investigations, all patients enrolled in the two arms ( study arm and control arm) of the study will be followed for one year (monthly visits for the first three months followed by visits three months until completion of study: total of 6 follow up visits) and the pre-specified investigations repeated at the one year follow up. In one arm (the control group), the patients will be offered best risk factor management strategies as currently being practiced by stroke specialists at HGH in Qatar. And in the second ( the subject group) arm, with assistance of a nurse-practitioner and pharmacist, the investigators will make aggressive attempts to meet "to target" defined risk factors and have the evaluations and investigations completed as in the initial year cohort. All patients will have risk factor stratification according the Framingham Risk Score (FRS) and the change in score measured over time.The primary objective will be to determine if an approach that utilizes a comprehensive strategy results in a significantly outcome. A clinically 'meaningful' difference in the blood pressure (BP) and lipid control of 10% between the aggressively managed versus patients treated with the standard of care will require minimum of 200 patients in each group (alpha error set at 0.05 and beta error at 0.20, power 80%) to be recruited over 1 year and followed for one year (total study duration 2 years).

All patients will have screening magnetic resonance imaging (MRI) (including gradient echo (GRE) sequence), carotid 3D Doppler measurement of plaque volume, and PAD assessments, C-reactive protein (CRP) and evaluation for protein urea at baseline. These studies will be repeated in 1 year at the time of exit from the study. The co-primary objective would be to monitor progression (or regression) of plaque build-up on 3D Doppler imaging of the carotid arteries between the two cohorts. The investigators hypothesize that aggressive management of vascular risk factors to "recommended target levels" will lead to better vascular health. Compared to current practice, comprehensive and coordinated approach at preventive measures will lead to more patients with better control of blood pressure and lipid levels. Improved risk factor management will result in slowing of atherosclerosis and its downstream effects which will be measurable on sophisticated blood and imaging testing. Clinically this will translate into fewer hospital re-admissions.

ELIGIBILITY:
Inclusion Criteria:

* ISCHEMIC STROKE OR TIA including ocular stroke such as Amaurosis Fugax, within the past year (not intracranial hemorrhage or due to trauma, malignancy or cardio-embolic related to structural heart disease)
* MEETS AT LEAST ONE OF THE FOLLOWING THREE CRITERIA:

  * systolic Bp>140 mmHg but <200 mmHg (at 24 HR from admission/if clinic visit 3 readings 5 minutes apart)
  * fasting LDL cholestrol >2.0 (MEASURED WITHIN PREVIOUS 6 MONTH)
  * total: HDL cholestrol ratio >4.0 (measured within previous 6 month)
* Willing to participate (by signing consent form)and willing to return for study-related scheduled follow up visits for one year from the time of enrollment into the study

Exclusion Criteria:

* Participation in concurrent interventional trial related to stroke or vascular disease
* Any condition, including foreshortened life-expectancy or severe comorbidities that would preclude treatment benefit or 12-month follow up.
* Institutionalized in a long term care facility
* Already on maximal therapy for risk factors:

  * On 3 ANTI HTN drugs at maximal dose (if htn is inclusion criteria)
  * On maximal dose of statin (if elevated LDL-cholesterol is inclusion criteria)
* CT or MRI shows evidence of primary intracranial hemorrhage or neoplasm
* Active coronary artery disease
* Severe Renal on hemo-dialysis(HD) or Severe Hepatic dysfunction
* Cognitive dysfunction severe enough to interfere with patients ability to give informed consent
* Severe systemic illness that will not allow for the patient to complete the one year trial
* History of intolerance to statins or commonly used anti-hypertensive medications(intolerance/contraindication to statin(if elevated LDL-c is the inclusion criteria)
* Unable to tolerate antiplatelet agents
* Decline of consent
* Reside outside Qatar
* Unable to participate (due cognition, mobility, language barrier)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2017-11-12 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression/regression of 3D plaque volume | one year
  3D carotid doppler imaging studies

SECONDARY OUTCOMES:
Measurement of blood pressure | one year
  management of life style
Measurement of Lipid levels | one year
  management of lifestyle

CONTACTS AND LOCATIONS:
Overall Officials: YAHIA Z BASHIER IMAM, MBBS,MRCP,MRCPE, Principal Investigator — Hamad Medical Corporation
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Imam YZ, Mohamed MFH, Abdelmoneim MS, Santos M, Alkhawad N, Salam A, Amir N, Saqqur M, Muhammad A, Elsoutohy A, Kamran S, Akhtar N, Kiliyanni AS, Own A, Deleu D, Shuaib A. Prospective study to optimize the health of patients with TIAS (transient ischemic attack) and stroke admitted to the Hamad General Hospital. Medicine (Baltimore). 2020 Jul 10;99(28):e20694. doi: 10.1097/MD.0000000000020694. PMID 32664066